CLINICAL TRIAL: NCT07310147
Title: Empower Your Mind to Embrace Your Life: Development and Efficacy Study of a Videoconference-delivered Group Intervention Based on Acceptance and Commitment Therapy for People With Young-onset Parkinson's Disease
Brief Title: Empower Your Mind to Embrace Your Life: an Online ACT Intervention for Young-Onset Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Inês Carolina Andrade Matos Pina, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.12842.BD
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD)
Keywords: Acceptance and Commitment Therapy; Parkinson's disease; Psychological Flexibility; Online group intervention
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This project will follow a longitudinal design. Individuals presenting a clinically established young-onset PD diagnosis will be allocated to the Control Group (no intervention; n ≥ 10) or to the Experimental Group (Empower your mind to embrace your life group intervention; n ≥ 10).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group of participants with young-onset diagnosis of Parkinson's disease (n ≥ 10) not subjected to any psychological intervention within the current study. Participants will be assessed at baseline, at post-intervention (immediately after session 8 of the intervention program), and at 3-month follow-up.
- Intervention Group (Experimental): Group of participants with young-onset diagnosis of Parkinson's disease (n ≥ 10) subjected to an 8-week online psychological intervention delivered in a group format (Empower your mind to embrace your life intervention). Participants in the experimental group will be assessed at baseline, post-intervention (immediately after session 8 of the intervention program), and at 3-month follow-up.
  Interventions: Behavioral: Empower your mind to embrace your life

INTERVENTIONS:
Behavioral: Empower your mind to embrace your life — An eight-session Acceptance and Commitment Therapy (ACT) for young-onset Parkinson's disease, applied in a group format and delivered online (via videoconferencing).
  Arms: Intervention Group

SUMMARY:
Parkinson's disease (PD) has a substantial impact on daily life and significantly affects functioning, mental health and quality of life. Although considered a disease of the elderly, an early diagnosis is also common. Non-pharmacological interventions have been increasingly recommended for PD, including psychotherapy, with emerging evidence suggesting that Acceptance and Commitment Therapy (ACT) may be suitable to support individuals living with PD. This project aims to expand the current evidence for ACT interventions in this population by developing, implementing, and investigating the preliminary efficacy of a novel online-delivered ACT intervention (Empower your mind to embrace your life) for individuals with a diagnosis of young-onset PD. For this purpose, a feasibility study will be conducted to assess the acceptability and preliminary efficacy of the intervention across two groups (control and ACT intervention). This group-based intervention consists of eight weekly sessions and will be delivered in an online format (via videoconferencing). Outcome measurement will be assessed at pre-intervention, post-intervention, and at 3-month follow-up. When comparing changes in outcome variables between the control and intervention groups at post-treatment, improvements are expected only in the intervention group. These improvements are also expected to be maintained over time (at 3-month follow-up). Lastly, changes in psychological (in)flexibility processes are expected to predict changes in outcome variables in the intervention group. This study will provide important insights to research and clinical practice by providing data on the feasibility and preliminary efficacy of this novel ACT-based intervention for the context of young-onset PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex, progressive neurodegenerative disease that predominantly affects movement. Although considered a disease of the elderly, an early diagnosis is also common and entails unique challenges that significantly affect several domains of life. PD is characterized by a multitude of motor (e.g., bradykinesia, resting tremor, rigidity) and non-motor symptoms (NMS, e.g., depression, pain, fatigue). Specifically, NMS have received increasing attention due to their detrimental impact on individuals' functioning, mental health outcomes and overall quality of life. In fact, NMS can be as disabling as motor PD manifestations, particularly in people with young-onset PD.

In recent years, non-pharmacological interventions have been developed with the aim of improving overall quality of life and managing NMS, including psychotherapy. In particular, third-wave psychological interventions have been applied in the context of PD with promising results, and literature has specifically highlighted Acceptance and Commitment Therapy (ACT) as a transdiagnostic model that appears to be well-suited for helping individuals with PD manage the challenges associated with their symptoms. The overarching goal of ACT is to increase psychological flexibility, a core process defined as the ability to be fully in contact with the present moment, with an accepting and nonjudgmental attitude, while behaving according to one's values. Evidence supports ACT's efficacy in several chronic physical illnesses, but few studies have implemented such interventions in adults diagnosed with PD. Despite promising results, current evidence remains limited and preliminary.

Additionally, literature highlighted the relevance of technology-supported psychological interventions in providing more cost-effective interventions for healthcare systems, especially in the context of chronic conditions. Notably, videoconferencing has been shown to be effective in overcoming face-to-face intervention-related barriers (e.g., mobility limitations, transport), which is particularly relevant in the context of PD.

Considering this background, the current project aims to contribute to the advance of ACT-based interventions in this field by developing, implementing, and examining the feasibility and preliminary efficacy of the "Empower your mind to embrace your life" intervention. This innovative ACT-based intervention was designed specifically to the context of young-onset PD and will be delivered online, in group format. The feasibility, acceptability and preliminary efficacy will be tested using a parallel-arm study, comparing the intervention with a control condition/waiting list (individuals with an early-onset PD diagnosis that will not receive any type of psychological intervention during the course of the study). Our hypothesis is that by targeting ACT core processes (e.g., acceptance, mindfulness, values), not only functioning and psychological outcomes will improve, but overall quality of life will be positively impacted. For this purpose, a longitudinal design will be implemented, including three assessment moments: baseline, post-intervention and 3-month follow-up (primary outcomes: health-related quality of life and psychopathology indicators -depression and anxiety symptoms; secondary outcomes: ACT core processes [chronic illness-specific and general psychological flexibility, chronic illness-related cognitive fusion, mindfulness], and other relevant outcomes, such as body functionality, shame). All procedures inherent to this research project were approved by the Ethics Committees of the Faculty of Psychology and Educational Sciences, University of Coimbra; Coimbra Local Health Unit (ULS Coimbra), and Hospital da Luz Coimbra. All participants provided their informed consent prior to data collection. The voluntary, confidential and pseudo-anonymized nature of the study was clearly explained. Participants were also informed about the option to decline participation or withdraw at any moment without any negative consequence. All participants will maintain their usual medical treatment, which includes medication for managing PD-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Young-onset PD diagnosis confirmed by a neurologist
* Classification between stages 1 and 2.5 according to the Hoehn &Yahr scale
* Aged between 21-65 years
* Fluent Portuguese speakers

Exclusion Criteria:

* Currently undergoing any form of psychology intervention
* Pregnancy
* Current suicidal ideation
* Diagnosis of severe psychiatric illness (e.g., severe depression, psychotic illness, bipolar disorder)
* Cognitive impairment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire - short form (PDQ-8) | Baseline, Week 8, 3-month follow-up
  The PDQ-8 was used to measure Parkinson's disease specific health-related quality of life through 8 items. This self-report instrument covers domains such as mobility, activities of daily living, emotional well-being, social support, communication, cognition, bodily discomfort and stigma. Each item is answered on a five-point Likert scale (ranging from 0 = Never; 4 = Always or cannot do at all). Higher scores on PDQ-8 represent poor health-related quality of life. Previous psychometric studies found very good internal consistency values. This measure was validated to the Portuguese population within the scope of this research project and showed good internal consistency.
Hospital Anxiety and Depression Scale (HADS) | Baseline, Week 8, 3-month follow-up
  The HADS is a self-report measure designed to assess the presence and severity of depressive and anxiety symptoms over the past week. This instrument comprises 14 items rated on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much or Most of the time). Higher scores indicate greater depression and anxiety symptomatology. The HADS presented good internal consistency in the original and in the Portuguese versions.

SECONDARY OUTCOMES:
Psy-Flex for Chronic Illness (Psy-Flex-CI) | Baseline, Week 8, 3-month follow-up
  The Psy-Flex-CI assesses chronic illness-related psychological flexibility through 6 items, each referring to one of the six core ACT processes. Participants were instructed to answer according to a 5-point Likert scale (1 = Almost never; 5 = Almost always). This self-report measure was developed and validated within the scope of this research project and presents good psychometric properties.
Multidimensional Psychological Flexibility Inventory - 24 (MPFI-24) | Baseline, Week 8, 3-month follow-up
  The MPFI-24 is a self-report measure that assesses psychological flexibility and inflexibility. The scale consists of 24 items answered on a 6-point Likert scale (ranging from 1 = Never true to 6 = Always true), referring to the last 2 weeks. The scores can be averaged to create a composite score representing global psychological flexibility and inflexibility, respectively. Previous psychometric information demonstrates adequate psychometric properties, including good internal consistency values.
Cognitive Fusion Questionnaire - Chronic Illness (CFQ-CI) | Baseline, Week 8, 3-month follow-up
  The CFQ-CI is a 7-item measure of cognitive fusion specifically related to the experience of having a chronic illness and its symptomatology. Items are rated on a 7-point Likert scale ranging from 1 (Never true) to 7 (Always true). CFQ-CI has demonstrated excellent internal reliability.
The Mindful Attention and Awareness Scale (MAAS) | Baseline, Week 8, 3-month follow-up
  The MAAS is a self-report measure of mindfulness at a trait-level, designed to assess attention and awareness of present moment daily activities. The scale consists of 15 items rated on a 6-point Likert scale (1 = Almost always; 6 = Almost never). Higher scores reflect greater dispositional mindfulness. This instrument has demonstrated good internal consistency.
External and Internal Shame Scale (EISS) | Baseline, Week 8, 3-month follow-up
  The EISS consists of 8 items that assess the experience of external ("Other people see me as not being up to their standards.") and internal ("I am different and inferior to others.") shame. Items are answered according to a 5-point Likert scale (0 = Never to 4 = Always), with higher scores indicating greater shame feelings. The scale presented good internal consistency.
Functionality Appreciation Scale (FAS) | Baseline, Week 8, 3-month follow-up
  This 7-item self-report scale evaluates functionality appreciation (e.g., "I appreciate my body for what it is capable of doing"). Items are answered in a 5- point Likert scale ranging from 0 (Never) to 5 (Always), with higher scores indicating greater body functionality appreciation. The scale presented good internal consistency.
The Work and Social Adjustment Scale (WSAS) | Baseline, Week 8, 3-month follow-up
  The WSAS is a 5-item measure of perceived functional impairment in daily activities that evaluate the extent of disease interference in several life areas (e.g., work, family, interpersonal relations, social and private leisure/hobbies activities, and home management). Items are answered on a 9-point scale (0 = not at all, 8 = severely). Higher scores reflect higher functional impairment. This instrument showed good internal consistency across several different health conditions.

OTHER OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | Baseline
  This brief questionnaire is a screening tool based on the DSM-IV criteria for major depressive disorder that assess the severity of depression symptoms (e.g., depressed mood, loss of interest, fatigue, and suicidal ideation). The scale consists of 9 items rated on a 4-point Likert scale (0 = Not at all, 3 = Nearly every day). The scale also comprises an additional item assessing the impact of symptoms on functioning (ranging from Not difficult at all to Extremely difficult). Higher scores indicate more severe depression symptoms. The scale showed good internal consistency.
Non-motor Symptoms Questionnaire (NMSQuest) | Baseline
  This instrument was designed to detect Parkinson's disease specific non-motor manifestations in several domains (e.g., depression and anxiety symptoms, cardiovascular, sexual function, sleep disorder) and comprises 30 items. Each item is answered according to a "yes" or "no" scale. Higher scores indicate higher frequency of non-motor manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Inês Matos-Pina, MSc, Principal Investigator — CINEICC - Center for Research in Neuropsychology and Cognitive Behavioral Intervention, Faculty of Psychology and Educational Sciences of the University of Coimbra; Cláudia Ferreira, PhD, Principal Investigator — CINEICC - Center for Research in Neuropsychology and Cognitive Behavioral Intervention, Faculty of Psychology and Educational Sciences of the University of Coimbra; Mariana Moura-Ramos, PhD, Principal Investigator — Unidade Local de Saúde de Coimbra (ULS Coimbra)
Locations (1):
- CINEICC, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared in accordance with data protection regulations.